CLINICAL TRIAL: NCT06419491
Title: Assisted Notification of Partners of Men Having Sex With Men Discovering Their Seropositivity
Acronym: NotiVIH
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ANRS, Emerging Infectious Diseases (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: ANRS95048
Record Dates: First submitted 2024-05-14; First posted 2024-05-17 (Actual); Last update posted 2024-05-23 (Actual); Status verified 2024-05

CONDITIONS: HIV Infections
Keywords: HIV; Partner notification tools
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Digital notification tool (No Intervention): A partner notification digital tool allowing the sending of anonymous or personalised standardised text messages to partners and an information leaflet are provided to index patients
- Digital notification tool and counseling (Experimental): In addition to the provision of the partner notification digital tool and the leaflet, a partner notification approach assisted by a trained counsellor during a specific counselling interview is offered to index patient.
  Interventions: Other: Partner notification by a trained counsellor

INTERVENTIONS:
Other: Partner notification by a trained counsellor — One (or more if needed) interview with a partner notification trained counsellor is offered to index patients. During the interview, the counsellor gives information on partner notification, helps the index patients to remember their partners, to assess their HIV/sexually transmitted infection exposure and explains options to notify them.
  During the interview, the index patient can choose to entrust the notification of some of their partners to the counsellor. However, according to French law, provider referral is permitted only when it is anonymous. Therefore, this option is reserved to partners with a lot of partners in order to limit the risk of identifying the index patient
  Arms: Digital notification tool and counseling

SUMMARY:
The context of HIV has changed dramatically this last two decades with the availability of highly active and well tolerated antiretroviral therapies, and the extension of prevention methods to include treatment as prevention of onward transmissions. It is time to test and treat as many HIV infected people as possible. HIV testing that target people known to have been exposed to HIV is an interesting option to explore to curb the spread of the epidemic. Notifying HIV exposed sexual partner for them to get an HIV test and treatment contribute to reduce HIV transmissions. The partner notification (PN) gives the opportunity to HIV positive partners to access to care and negative partners, access to prevention services.

Several tools have been developed worldwide, in particular in the United Kingdom and the US, to help HIV or index patients to notify their sexual partner or needle-sharing people. This approach is new in France and PN intervention has to be assessed.

The present study aimed to assess the effectiveness of a digital PN tool or a counselling interview to help men having sex with men (MSM) newly diagnosed for HIV to notify their exposed partners. The study also aimed to evaluate the acceptability of these PN intervention in index patients and their notified partners in the French context.

To meet the objectives, an interventional study was developed in index patients (described above) coupled with :

* an observational study in notified partners to assess their PN acceptability and their HIV testing uptake after being notified
* a qualitative study in a sample of index patients and notified partner to assess more in depth their PN acceptability.

Expected results and perspectives Feasible and effective, assisted PN services may complete HIV testing offer (and by extension sexually transmitted infections screening) as well as the prevention offer Pre-Exposure Prophylaxis (PrEP) for MSM.

The study will provide information enabling the best practice guides. In a next step, PN interventions adapted to other key populations will be studied.

DETAILED DESCRIPTION:
Interventional study (supplementary information)

This is a cluster-randomised interventional study that will compare two interventional arms:

* The provision of a partner notification (PN) digital tool allowing the sending of anonymous or personalised standardised text messages to partners (Tool arm).
* In addition to the provision of the PN digital tool, a PN approach assisted by a counsellor during a specific counselling interview and the option for the index patient to entrust the notification of some of their partners to the counsellor (Tool + Counselling arm). Notification of partners by the counsellor should be anonymous and reserved for partners for whom the risk of re-identification of the index case is very low.

Randomisation of the centres 1:1.

The PN intervention will be offered to index patients at the time of HIV diagnosis or antiretroviral treatment initiation. They will have the option to use the available tools and to notify all or some of their partners.

Data on participant profile, PN assessment, acceptability, and consequences are collected by online self-administered questionnaires on a secure website. The one on participants' profile is available at enrollment and the another that collect the PN experience, one month later. The participant is invited by email to connect on the website and fill in the questionnaires.

The calculation of the number of index patients was based on the main outcome: increase the number of notified partners.

Considering a difference between the two arms of 34%, statistical power of 80%, risk of 5% and intra-cluster coefficient correlation of 0,03 with one-way test, 1104 exposed partners have to be stated in each arm. In median, MSM had 7 sexual partners within the 6 months before HIV diagnosis, ie. 157 index patients per arm.

This number was rounded to 200 index patients per arm to take into account uncertainty about de the correlation coefficient and enable analysis adjusted for 6 confusion factors.

Observational study in notified partners The PN message, delivered either through the digital tool or paper cards, informs the partners about their HIV/sexually transmitted infection (STI) exposure and invites them to get tested. It also contains a link to a website with information on PN, HIV testing and an invitation to participate in this study as a notified partner.

The objectives of this part are to:

* assess the HIV testing uptake after notification
* estimate the HIV positivity rate among notified partners
* describe the PN experience
* evaluate the acceptability of notified partners, whatever they get or not HIV testing

Notified partner register themselves on the study website. Like index patients, data on participant profile, PN acceptability, HIV testing and according to the test result, the linkage to care or to Pre-Exposure Prophylaxis (PrEP) are collected by online self-administered questionnaires on a secure website. The one on participants' profile is available at enrollment and the another that collect the PN experience and HIV testing, one month later. The participant is invited by email to connect on the website and fill in the questionnaires.

Qualitative study A qualitative study based on individual interviews will be conducted with a sample of participants (index patients and notified partners) to assess more in depth the acceptability of HIV PN, identify the barriers and levers of PN, as well as the components of intervention in the PN process that need to be adapt. Around 30 interviews will be conducted according to the principle of data saturation.

ELIGIBILITY:
Inclusion Criteria:

* men
* aged ≥18
* having sex with ≥2 men in the last 12 months
* diagnosed for HIV since ≤3 months at the time of inclusion

Exclusion criteria:

* Persons who do not provide an email address, needed to receive the study questionnaires
* Persons who do not speak or read French
* Persons subject to a legal protection measure (guardianship, safeguard of justice)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
The percentage of partners notified one month after the intervention, among the number of exposed partners stated by index patients | One month after the intervention
  An emailed invitation to complete an online self-administered questionnaire will be send to index patients to carry out an assessment of the notification process (number of partners exposed, contacted, notified, etc). Up to 3 reminders will be sent if no response.

SECONDARY OUTCOMES:
Percentage of acceptability of partner notification by index patients | One month after the intervention
  Percentage of index patients who notified at least one exposed partner
Percentage of adverse events of partner notification reported by index patients | One month after the intervention
  Percentage of index patients who reported violence, social harm, feeling left out from sexual partners.

CONTACTS AND LOCATIONS:
Overall Officials: Jade Ghosn, MD PhD, Study Director — AP-HP Hôpital Bichat Claude-Bernard, Paris, France